CLINICAL TRIAL: NCT01903096
Title: A Pilot Study to Treat Emotional Disorders in Primary Care With Evidence-based Psychological Techniques: A Randomized Controlled Trial
Brief Title: Treating Emotional Disorders in Primary Care With Psychological Techniques
Acronym: PsychPC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Psicofundación: Fundación Española para Promoción, Desarrollo Científico y Profesional de la Psicolo (Other)
Collaborators: Ministry of Health, Spain (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AP105162012; 2013-001955-11 (EudraCT Number)
Record Dates: First submitted 2013-07-02; First posted 2013-07-19 (Estimated); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Anxiety Disorders; Mood Disorders; Somatization Disorder; Pain Disorder
Keywords: Panic disorder; Generalized anxiety disorder; Social phobia; Specific phobia; Major depressive disorder; Dysthymia; Somatizations disorder; Pain disorder
MeSH Terms: conditions — Anxiety Disorders; Mood Disorders; Somatoform Disorders; Panic Disorder; Generalized Anxiety Disorder; Phobia, Social; Phobia, Specific; Depressive Disorder, Major; Dysthymic Disorder | interventions — Antidepressive Agents; Sleep; Acetaminophen

STUDY DESIGN:
Intervention Model Description: Randomised, controlled, two arm single-blind trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: A computer-generated allocation sequence was used to randomly assign patients (1:1) to receive either TD-GCBT plus TAU or TAU alone. All patients were assigned a code for blinding purposes and then the patient characteristics were sent to one of the investigators to check that they met the inclusion criteria. Patients who met the inclusion criteria were then randomized as described above.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive Behavioral Treatment (CBT) (Experimental): Cognitive Behavioral Treatment. Seven 90-minute sessions of group treatment along 24 weeks.
  Interventions: Behavioral: Cognitive Behavioral Treatment
- Treatment-As-Usual (TAU) (Active Comparator): Primary Care Treatment As Usual
  Interventions: Drug: Primary Care Treatment As Usual

INTERVENTIONS:
Behavioral: Cognitive Behavioral Treatment — Seven ninety-minute sessions of evidence-based psychological techniques designed to treat anxiety, depression and somatization disorders during a period of 24 weeks.
  Other Names: CBT (Cognitive-Behavioral Treatment)
  Arms: Cognitive Behavioral Treatment (CBT)
Drug: Primary Care Treatment As Usual — Usual treatment offered in Primary Care Services: depending on the diagnoses, patients will be prescribed different medications until symptoms disappear.
  Other Names: Antidepressants, antianxiety, sleep and pain medication.
  Arms: Treatment-As-Usual (TAU)

SUMMARY:
The strong demand for primary care (PC) services in Spain exceeds resources. Part of this demand is due to the increasing number of anxiety, depression, and somatization disorders that affect the general population. These disorders, commonly known as emotional disorders, are very common in Spanish PC settings, they are poorly detected by physicians, rarely receive adequate treatment (if they receive treatment it is mostly drugs instead of psychological treatment), they generate a highly frequent use of PC services, a greater burden than physical diseases and tend to become chronic without treatment.

Other countries have successfully put psychological techniques in PC into practice (in the United Kingdom the program known as "Improving Access to Psychological Therapies" has obtained very positive results) in order to correctly diagnose and treat emotional disorders. The results obtained in terms of symptoms, quality of life, diagnosis, etc., have been better than the usual treatment offered in PC services, involving no side effects, fewer relapses, and lower costs in the long term.

The general aim of this study is to test how well a psychological treatment program for anxiety, depression, and somatization disorders works in PC and to compare the results obtained after seven 90-minute group sessions (every to two to four weeks approximately, for a period of 24 weeks) with the usual treatment offered in Spanish PC services. Similar results to the ones already obtained in other countries are expected to be found.

Approximately 1130 adults, regardless of their age and sex, with an anxiety, depression and/or somatization disorder (diagnosed with a simple and short questionnaire) will participate in this study.

Participation will be voluntary and confidentiality will be guaranteed. Half of the participants in the study will be randomly assigned to receive their usual care and the other half will receive psychological treatment, within the same health care centre. Since it is a "double-blind" study, neither the health professional nor the patient will know which treatment will be applied. Psychological assessments will be carried out before and after receiving treatment and participants will be followed up at 3, 6 and 12 months.

Participation will pose no risks different from the typically present when receiving usual treatment. The aim of this study will be to maximize benefits and reduce potential harms (principle of proportionality).

DETAILED DESCRIPTION:
Secondary objectives:

* The experimental in comparison with the control group will report a greater decrease (including pre-post-treatment differences and follow-up at 3, 6 and 12 months) in emotional symptoms (total scores of anxiety, depressive and somatic symptoms as measured by the Patient Health Questionnaire), cognitive factors, and percentage of cases with probable emotional disorders (anxiety, depression, and somatization disorders).
* The experimental in comparison with the control group will report a decrease in its levels of work, family and social impairment (Sheehan Disability Scale), and an increase in its levels of physical health, psychological, social, and environmental quality of life (as measured by the different World Health Organization Quality of Life; WHOQOL-BREF scales).
* The experimental group in comparison with the control group will reduce the frequency of Primary Care visits (as well as other health care costs) at 6 month follow-up.
* In addition, the experimental group will report higher treatment satisfaction than the control group.

The following variables will be assessed:

* Clinical symptoms (anxiety, depression, somatizations), levels of adjustment (work, family, social),
* Quality of life (physical health, psychological, social, environmental),
* Emotional symptoms and thoughts (worries, beliefs, coping strategies, negative thoughts, etc.),
* Treatment satisfaction
* Frequent use of services
* Psychoactive drug use.

Patient recruitment

Inclusion criteria:

• Any adult patient seeking Primary Care treatment at any of the selected sites in Spain with a probable anxiety, mood and/or somatisation disorder (diagnosed with the Patient Health Questionnaire; PHQ-9) may voluntarily participate in the study regardless of his/her age and sex.

Exclusion criteria:

* Patients with severe mental disorders (e.g., bipolar disorder, personality disorder)
* Patients with a history of frequent or recent suicide attempt(s)
* Patients with a high level of disability (as measured by the Sheehan Disability Scale) who seek Primary Care treatment.
* Patients with severe anxiety disorders (e.g., comorbid substance use disorders) and severe mood disorders (Patient Health Questionnaire; PHQ-9 total score >= 20).
* Patients who do not meet diagnostic criteria for a probable emotional disorder or do not reach the established Patient Health Questionnaire cut-off points.

The minimum sample size required to obtain a significant result has been calculated with the Sample-Power SPSS program. The study should include 563 patients in each condition, with a total of 1126 patients, accounting for a 20% attrition or dropout. With this sample size, the result will be statistically significant (85% statistical power) when comparing both groups, even if they differ by one point only, with a standard deviation of 5, a range of scores from 0-27 for the PHQ-9, and it will enable us to conclude that the result is different for each group with a 95% confidence level.

Both groups will be equivalent in all measures before receiving treatment. 2x2 within and between-groups analyses of variance (group x treatment) will be conducted for each dependent variable. The effect size for each dependent variable will be calculated in both groups, as well as the 95% confidence interval, taking into account the number of treatment sessions. Primary analyses will follow the "intention-to-treat" principle in such a way that all individuals who participate in the study will be considered as members of one group even if they have not yet completed the protocol. "Therapeutic success" will be obtained if the average scores of the experimental group are significantly lower than those of the control group in the dependent variables (anxiety, depression, and somatization symptoms), and when the effect sizes are medium to large and significantly higher than those of the control group (especially in the case of anxiety symptoms). In addition, the results obtained by each group in terms of degree of disability (work, family and social), quality of life, treatment satisfaction, costs and cost-efficiency of both treatments will be compared.

It will be carried out in twenty five Primary Care (PC) centres in Madrid, Valencia, Albacete, Mallorca, Murcia, Vizcaya, Cordoba, Galicia, and Cantabria, and may be extended to other centres and cities.

It is expected to start in September 2013 and posttreatment will end by December 2018. The study will be open to participants until recruitment is completed. The follow-up period will end by September 2019.

Psicofundación (Spanish Foundation for the Promotion, Scientific and Professional Development of Psychology) and the Spanish Ministry of Economy and Competitiveness are funding this three-year project.

The main contact is Dr. Antonio Cano-Vindel, professor at the Faculty of Psychology of Complutense University of Madrid. E-mail: canovindel@psi.ucm.es. Telephone: (34)607705740.

ELIGIBILITY:
Inclusion Criteria:

* Any adult patient seeking Primary Care treatment at any of the selected sites in Spain with a probable anxiety, mood and/or somatisation disorder (diagnosed with the Patient Health Questionnaire) may voluntarily participate in the study regardless of his/her age and sex.

Exclusion Criteria:

* Patients with severe mental disorders (e.g., bipolar disorder, personality disorder)
* Patients with a history of frequent or recent suicide attempt(s)
* Patients with a high level of disability (as measured by the Sheehan Disability Scale) who seek Primary Care treatment.
* Patients with severe anxiety disorders (e.g., comorbid substance use disorders) and severe mood disorders (Patient Health Questionnaire; PHQ-9 total score >= 20).
* Patients who do not meet diagnostic criteria for a probable emotional disorder or do not reach the established PHQ cut-off points.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1126 (Actual)
Dates: Start 2014-01-14 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Anxiety symptoms after psychological treatment versus Primary Care usual treatment. | Up to two years
  Diagnostic and Statistical Manual of Mental Disorders -Fourth Edition (DSM-IV) clinical symptoms of anxiety (total frequency scores in anxiety as measured by the Patient Health Questionnaire) as reported by patients after receiving psychological treatment or usual treatment.
Depressive symptoms after psychological treatment versus Primary Care usual treatment. | Up to two years.
  Diagnostic and Statistical Manual of Mental Disorders -Fourth Edition (DSM-IV) clinical symptoms of depression (total frequency scores in depression as measured by the Patient Health Questionnaire) as reported by patients after receiving psychological treatment or usual treatment.
Somatic symptoms after psychological treatment versus Primary Care usual treatment. | Up to two years.
  Diagnostic and Statistical Manual of Mental Disorders -Fourth Edition (DSM-IV) somatic symptoms (total frequency scores in somatic symptoms as measured by the Patient Health Questionnaire) as reported by patients after receiving psychological treatment or usual treatment.

SECONDARY OUTCOMES:
Cognitive factors after psychological treatment versus Primary Care usual treatment. | Up to two years
  Pre-post treatment differences at post treatment and at 3, 6 and 12 month follow-up in cognitive tests scores (composite score designed to assess ruminative processes, pathological worry, attentional and interpretive biases, emotion regulation strategies and metacognitive beliefs) as reported by patients after receiving psychological treatment or usual treatment.
Level of impairment after psychological treatment versus Primary Care usual treatment. | Up to two years
  Pre-post treatment differences at post treatment and at 3, 6 and 12 month follow-up in work, family and social impairment (as measured by the Sheehan Disability Scale) as reported by patients after receiving psychological treatment or usual treatment.
Quality of life after psychological treatment versus Primary Care usual treatment. | Up to two years
  Pre-post treatment differences at post treatment and at 3, 6 and 12 month follow-up in physical health, psychological, social, and environmental quality of life (as measured by the different World Health Organization Quality of Life; WHOQOL-BREF scales) as reported by patients after receiving psychological treatment or usual treatment.
Frequency of primary care visits after psychological treatment versus Primary Care usual treatment. | Up to 18 months
  Frequency of primary care visits after psychological treatment versus Primary Care usual treatment.

OTHER OUTCOMES:
Treatment satisfaction | Up to 18 months
  Treatment satisfaction after receiving psychological treatment versus treatment as usual.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio R Cano-Vindel, Professor, Study Director — Universidad Complutense de Madrid
Locations (1):
- Complutense University of Madrid, Madrid, Spain

REFERENCES:
- [Background] Cano-Vindel A. Los desórdenes emocionales en Atención Primaria [Emotional Disorders in Primary Care]. Ansiedad y Estrés 2011;17(1):73-95.
- [Background] Cano-Vindel A; Wood CM; Dongil E; Latorre JM. El trastorno de pánico en Atención Primaria [Panic disorder in Primary Care]. Papeles del Psicólogo 2011;32(3):3-13.
- [Background] Cano-Vindel A. Bases teóricas y apoyo empírico de la intervención psicológica sobre los desórdenes emocionales en Atención Primaria. Una actualización [Theoretical and empirical evidence supporting a psychological intervention for emotional disorders in Primary Care. An update]. Ansiedad y Estrés 2011;17(2-3):157-184.
- [Background] Cano-Vindel A; Dongil-Collado E; Salguero JM; Wood CM. Intervención cognitivo-conductual en los trastornos de ansiedad: una actualización [Cognitive-behavioral treatment for anxiety disorders: an update]. Informació Psicològica 2011;102:4-27.
- See also: Spanish Society for the Investigation of Anxiety and Stress — http://www.ansiedadyestres.org/